CLINICAL TRIAL: NCT03451747
Title: The Potential Role of Testosterone Between Hypertension and Target Organ Damage in Postmenopausal Hypertensive Women
Brief Title: The Potential Role of Testosterone on Target Organ Damage in Postmenopausal Hypertensive Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Jing Yu, Principal Investigator, LanZhou University
Other Study IDs: LanZhou
Record Dates: First submitted 2018-02-18; First posted 2018-03-02 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
Keywords: hypertension; female
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- postmenopausal hypertensive women
- mached hypertensive men

SUMMARY:
The incidence of CVD-related deaths is generally higher in women than men. Postmenopausal changes in estrogen/androgen ratio that induce a relative androgen excess have been proposed as important factors in the higher prevalence of hypertension. Therefore, the investigators hypothesize that testosterone has potential role between hypertension and target organ damage in postmenopausal hypertensive women. And the objective is to evaluate the effects of testosterone between hypertension and target organ damage in postmenopausal hypertensive women.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension
* Women are all postmenopausal
* Men are matched with women.

Exclusion Criteria:

* Secondary hypertension
* Coronary disease
* Heart failure
* Arterial fibrillation
* Previous myocardial infarction
* Previous stroke
* Malignant disease
* Kidney failure
* Liver failure
* Neoplastic disease
* Severe neurological diseases
* Severe metabolic or organic decompensation
* Refuse to sign the informed consent form

Ages: 45 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 322 hypertensive patients hospitalized in our department from 2016 to 2017 were enrolled. Included 161 postmenopausal hypertensive women and 161 mached hypertensive men.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2018-03-10 (Estimated); Primary Completion 2018-04-05 (Estimated); Study Completion 2018-04-05 (Estimated)

PRIMARY OUTCOMES:
Relative indexes of myocardial remodeling | Baseline
  Cardiac structure (left ventricular mass index in grams for square meter) measurement.
Ambulatory blood pressure monitoring | Baseline
  Non-invasive ambulatory blood pressure monitoring (ABPM) was performed for every enrolled patient with an ABPM equipment.
The level of testosterone (T) | Baseline
  Blood samples used to analyze the levels of sexual hormones were collected between morning 8:00 and 9:00 after an overnight fast. Testosterone (T) units on nanogram per deciliter.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang S, Yu H, Jing C, Liang W, Chen L, Lin Y, Li R, Yu J, Li N. Correlation between ambulatory blood pressure indices and sex hormone imbalance in hypertensive women with different menopausal durations: a cross-sectional study. Eur J Med Res. 2026 Jan 19;31(1):95. doi: 10.1186/s40001-025-03797-5. PMID 41555389
- [Derived] Li N, Ma R, Wang S, Zhao Y, Wang P, Yang Z, Jin L, Zhang P, Ding H, Bai F, Yu J. The potential role of testosterone in hypertension and target organ damage in hypertensive postmenopausal women. Clin Interv Aging. 2019 Apr 29;14:743-752. doi: 10.2147/CIA.S195498. eCollection 2019. PMID 31118595